CLINICAL TRIAL: NCT04281901
Title: Efficacy of Platelet- and Extracellular Vesicle-rich Plasma for the Treatment of Chronically Inflamed Post-surgical Temporal Bone Cavities: a Randomised Controlled Clinical Study
Brief Title: Efficacy of Platelet- and Extracellular Vesicle-rich Plasma in Chronic Postsurgical Temporal Bone Inflammations
Acronym: PvRP-ear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other); University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Domen Vozel, MD, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0120-146/2019/5
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Results first posted 2020-08-13 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Otitis Media Chronic; Temporal Bone
Keywords: Otitis Media; Mastoidectomy; Wound Healing; Platelet-Rich Plasma; Extracellular Vesicles; Cholesteatoma; Regenerative Medicine
MeSH Terms: conditions — Otitis Media; Cholesteatoma | interventions — Platelet Count

STUDY DESIGN:
Intervention Model Description: Participants treated with PVRP will receive PVRP-soaked ear wicks at the day of recruitment, additionally 1 month later and then followed-up twice in 1-month intervals. Participants not treated with PVRP will be treated with standard conservative nonsurgical measures with the same follow-up time.
Who Masked: Outcomes Assessor
Masking Description: A person unaware of the participants and their random allocation will measure inflammation area with computer software provided by ZEN Lite, Zeiss.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVRP treated participants (Experimental): Participants will receive PVRP in the chronically inflamed radical cavity at the baseline evaluation (day 0) and 1 month later (1. follow-up). There will be 2 additional follow-ups with a 1-month interval.
  Interventions: Drug: Platelet- and extracellular vesicle-rich plasma
- Standardly treated participants (Active Comparator): Participants will receive standard conservative measures for the chronically inflamed radical cavity at the baseline evaluation (day 0), 1 month later (1. follow-up), 2 months later (2. follow-up) and 3 months later (3. follow-up).
  Interventions: Drug: Standard conservative treatment

INTERVENTIONS:
Drug: Platelet- and extracellular vesicle-rich plasma — ear wick soaked in platelet- and extracellular vesicle-rich plasma
  Arms: PVRP treated participants
Drug: Standard conservative treatment — standard conservative measures, including antimicrobials, antiseptics and aural toilette for treating a chronically inflamed radical cavity.
  Arms: Standardly treated participants

SUMMARY:
This clinical study evaluates the efficacy of the autologous blood-derived product called platelet- and extracellular vesicle-rich plasma (PVRP) for the treatment of chronically inflamed post-surgical temporal bone cavities. Half of the participants will be treated with platelet- and extracellular vesicle-rich plasma and another half with standard nonsurgical measures.

DETAILED DESCRIPTION:
The hypothesis of this study is that platelet- and extracellular vesicle-rich plasma (PVRP) may be efficient in the treatment of chronically inflamed post-surgical temporal bone cavities.

Platelet-rich plasma (PRP) is a well-known autologous blood-derived product with favourable immune, haemostatic and regenerative effects. It has been used in various medical fields including otorhinolaryngology.

In fact, PRP contains important concentrations of extracellular vesicles (EV) which are the main contributors to PRP effects. For that reason, PRP can be identified as platelet- and extracellular vesicle-rich plasma (PVRP). In this study, PVRP will be prepared by a unique non-commercial 2-step centrifugation protocol developed by this study researchers.

A radical cavity is a large post-surgical temporal bone cavity due to removal of the posterior external ear canal wall in open-technique cholesteatoma surgery. This technique is performed in approximately 40 per cent of cholesteatoma surgery.

Radical cavities become inflamed in 3-20 per cent, which leads to the formation of granulation tissue and multiple suppurative periods. The large spectrum of surgical and nonsurgical treatment options have been applied to reduce patient discomfort. This significantly worsens the patients' quality of life and puts a significant burden on health care.

Due to the knowledge of local immune response mechanisms in moist radical cavities and exhausted treatment options, new conservative treatment options have been researched. PVRP could present a promising treatment option for chronically inflamed radical cavities based on published preclinical and clinical studies.

PVRP will be administered to chronically inflamed radical cavities via PVRP-soaked ear wicks.

ELIGIBILITY:
Inclusion Criteria:

* chronic otitis media, defined as a presence of at least 1 of the following: visible ear discharge, indirect signs of ear discharge (e.g. on a pillow, clothes), ear itching, the sensation of ear fullness, clinical signs of acute exacerbation of chronic otitis media during an otomicroscopic examination.
* non-cholesteatomatous chronic otitis media despite prior standard conservative treatment
* non-cholesteatomatous chronic otitis media despite prior surgical treatment

Exclusion Criteria:

* the presence or suspicion of cholesteatoma
* infection of venepuncture site
* pregnancy
* breastfeeding
* long-term treatment with antimicrobial drugs
* long-term treatment with immunosuppressant drugs
* the presence of systemic infectious disease
* the presence of an autoimmune disease
* the presence of cancer
* receiving other types of experimental treatment for chronic otitis media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saba Battelino, MD, PhD, Study Chair — Department of Otorhinolaryngology and Cervicofacial Surgery, UMC Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
IPD relevant for the results will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from the beginning of the study until the conclusion.
Access Criteria: Access for the data affecting results will be provided. Access to this data will be provided by the central contact person or central contact backup. No personal identification information will be provided.

REFERENCES:
- [Background] Vozel D, Ursic B, Krek JL, Stukelj R, Kralj-Iglic V. Applicability of extracellular vesicles in clinical studies. Eur J Clin Invest. 2017 Apr;47(4):305-313. doi: 10.1111/eci.12733. Epub 2017 Feb 28. PMID 28156006
- [Background] Uršič B, Vozel D, Šuštar V, Kocjančič B, Dolinar D, Kralj-Iglič V. Extracellular Vesicles from Platelet-Rich Plasma as Conveyors of Regeneration Potential in Orthopedics. J Hematol Thromboembolic Dis 2(5), 2014.
- [Result] Vozel D, Bozic D, Jeran M, Jan Z, Pajnic M, Paden L, Steiner N, Kralj-Iglic V, Battelino S. Autologous Platelet- and Extracellular Vesicle-Rich Plasma Is an Effective Treatment Modality for Chronic Postoperative Temporal Bone Cavity Inflammation: Randomized Controlled Clinical Trial. Front Bioeng Biotechnol. 2021 Jul 7;9:677541. doi: 10.3389/fbioe.2021.677541. eCollection 2021. PMID 34307321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 participants with chronic postoperative temporal bone cavity inflammation were recruited at the tertiary otorhinolaryngology referral centre between February- March 2020. In this period the list of patients was created based on examinations and documentation review. 2 participants had bilateral involvement, therefore 27 cases were recruited.
Pre-assignment Details: After random allocation 1 patient allocated to the group treated with standard conservative measures refused to participate in the study.
Units Other Than Participants: case
Groups:
- PVRP Treated Participants: Participants received platelet- and extracellular vesicle-rich plasma (PVRP)-soaked ear wick in the chronic postoperative temporal bone cavity inflammation at the baseline evaluation (i.e., 1. check-up) and 1 month later (i.e., 2. check-up). Two additional check-ups were performed in a 1-month interval. The aural toilet was applied at each check-up. No other treatment measures were applied
  Platelet- and extracellular vesicle-rich plasma: ear wick soaked in platelet- and extracellular vesicle-rich plasma
- Standardly Treated Participants: Participants were treated with standard conservative measures, including antimicrobials, antiseptics and aural toilette at 1., 2., 3. and 4. check-up.
  Standard conservative treatment: standard conservative measures, including antimicrobials, antiseptics and aural toilette for treating a chronically inflamed radical cavity.
Period: Overall Study
Arm/Group | PVRP Treated Participants | Standardly Treated Participants
Started (Baseline evaluation (i.e., first check-up)) | 12; 12 case | 12; 14 case
2. Check-up (1 month after the baseline evaluation) | 11; 11 case | 11; 13 case
3. Check-up (2 months after baseline evaluation) | 11; 11 case | 11; 13 case
Completed (4. check-up (i.e., 3. months after the baseline evaluation)) | 11; 11 case | 11; 13 case
Not Completed | 1; 1 case | 1; 1 case

BASELINE CHARACTERISTICS:
Units Other Than Participants: case
Groups:
- Total: Total of all reporting groups
Arm/Group | PVRP Treated Participants | Standardly Treated Participants | Total
Number analyzed (Participants) | 11 | 11 | 22
Number analyzed (case) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (18) | 52 (24) | 50 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Slovenia | 11 | 11 | 22
Quality of life (i.e., COMQ-12 sum score) [Mean (Standard Deviation); unit: scores on a scale] — Quality of life, related to chronic postoperative temporal bone cavity inflammation was measured with Slovenian version of COMQ-12 (Chronic Otitis Media Questionnaire-12). The questionnaire consists of 12 questions, scored 0-5. The higher sum score signifies the worse quality of life. The minimum sum score is 0 and the maximum is 60.
  scores on a scale | 32 (10) | 31 (10) | 31 (10)
Presence of bacteria in temporal bone cavity [Count of Units; unit: case] — Bacteria were identified in the temporal bone cavity by microbiological examinations of temporal bone cavity swabs.
  case
    Bacteria identified | 10 | 12 | 22
    Bacteria not identified | 1 | 1 | 2
Presence of fungi in temporal bone cavity [Count of Units; unit: case] — Fungi were identified in the temporal bone cavity by microbiological examinations of temporal bone cavity swabs.
  case
    Fungi identified | 2 | 3 | 5
    Fungi not identified | 9 | 10 | 19
Comorbidities [Count of Participants; unit: Participants]
  Comorbidities present | 6 | 6 | 12
  Comorbidities absent | 5 | 5 | 10
Allergies [Count of Participants; unit: Participants]
  Allergies present | 5 | 4 | 9
  Allergies absent | 6 | 7 | 13
Regular medications [Count of Participants; unit: Participants] — Presence or absence of regular medication intake.
  Participants
    Intake of regular medications | 3 | 6 | 9
    No intake of regular medications | 8 | 5 | 13
Coagulopathy [Count of Participants; unit: Participants] — Presence of coagulopathies, including medication-related coagulopathies.
  Participants
    Presence of coagulopathy | 2 | 1 | 3
    Absence of coagulopathy | 9 | 10 | 19
Smoking [Count of Participants; unit: Participants]
  Smoking | 2 | 5 | 7
  Not smoking | 9 | 6 | 15
Alcohol intake [Count of Participants; unit: Participants]
  Regular alcohol intake | 10 | 7 | 17
  No regular alcohol intake | 1 | 4 | 5
Time to treatment according to the study protocol [Median (Full Range); unit: years] — Time to treatment according to the study protocol refers to the time from the beginning of the complaints due to the chronic postoperative temporal bone cavity inflammation to the baseline evaluation.
  years | 7.4 [0.2 to 9.0] | 8.7 [0.7 to 9.2] | 8.1 [0.2 to 9.2]
Time from otosurgery to treatment according to the study protocol [Median (Full Range); unit: years] — Time from otosurgery refers to the time from the last otological surgical procedure (i.e., due to the temporal bone disease which led to the chronic postoperative temporal bone cavity inflammation) to the baseline evaluation. Population: Data of time from otosurgery was unknown some cases.
  years
    number analyzed (case) | 10 | 8 | 18
    (all) | 12.7 [0.5 to 59.1] | 14.3 [3.0 to 34.9] | 13.8 [0.5 to 59.1]
Underlying otological disease requiring otosurgical treatment [Count of Units; unit: case]
  Middle ear cholesteatoma | 10 | 12 | 22
  External auditory canal squamous cell-carcinoma | 0 | 1 | 1
  External auditory canal cholesteatoma | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammation Surface Area.
Description: The inflamed tissue in the postoperative temporal bone cavity was observed and photographed otomicroscopically. Then the surface area of the inflamed tissue was determined by using ZEN 3.0 blue edition software(©Carl Zeiss Microscopy GmbH, 2019).
  Values in square millimetres were transformed to the ratios of the inflamed surface area according to the baseline surface area. The baseline surface area values are therefore 100% for each case or participant.
Time Frame: Baseline, 1 month, 2 months and 3 months after baseline
Measure: Mean (Standard Deviation); unit: percentage of the baseline surface
Units Other Than Participants: case
Arm/Group | PVRP Treated Participants | Standardly Treated Participants
Number analyzed (Participants) | 11 | 11
Number analyzed (case) | 11 | 13
percentage of the baseline surface
  Baseline evaluation | 100 (0) | 100 (0)
  1 month | 43 (30) | 135 (35)
  2 months | 36 (30) | 144 (64)
  3 months | 36 (28) | 150 (97)

2. Primary Outcome: Change in Chronic Otitis Media Questionnaire 12 Score
Description: Sum score of Chronic Otitis Media Questionnaire 12 (COMQ-12), patient-reported health-related quality of life measure.
  Each question is scored from 0 to 5 points, therefore the minimum score value is 0 and the maximum 60.
  A higher score means worse chronic otitis media-related quality of life. A higher change in COMQ-12 score means a better treatment outcome.
Time Frame: Baseline, 1 month, 2 months and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PVRP Treated Participants | Standardly Treated Participants
Number analyzed (Participants) | 11 | 11
score on a scale
  baseline evaluation (i.e., 1. check-up) | 32 (10) | 31 (10)
  2. check-up | 22 (12) | 34 (10)
  3. check-up | 20 (11) | 33 (11)
  4. check-up | 17 (10) | 32 (8)

3. Secondary Outcome: Bacterial Presence
Description: The microbiological analysis included incubation of smear samples to cultivate bacteria, present in postsurgical temporal bone cavity inflammation. Microscopical analyses of colonies were performed to identify the presence of bacteria. Bacteria were absent if no colonies were identified.
Time Frame: Baseline, 2 months
Measure: Count of Units; unit: case
Units Other Than Participants: case
Arm/Group | PVRP Treated Participants | Standardly Treated Participants
Number analyzed (Participants) | 11 | 11
Number analyzed (case) | 11 | 13
case
  bacteria identified at the 2. check-up | 7 | 9
  bacteria not identified at the 2. check-up | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the beginning of the trial to the last check-up, i.e. from the baseline evaluation and 4 months after (4. check-up). Therefore, the adverse effects were monitored for 4 months.
Description: 11 patients who received platelet- and extracellular vesicle-rich plasma (PVRP) and 11 who received standard conservative treatment measures were at risk for serious adverse events, all-cause mortality and other adverse events. PVRP-related adverse events were defined as worsening of chronic postsurgical temporal bone inflammation due to PVRP. The worsening was attributed to PVRP if worsening of the clinical picture occurred within three days after PVRP administration.
Arm/Group | PVRP Treated Participants | Standardly Treated Participants
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04281901/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04281901/SAP_001.pdf